CLINICAL TRIAL: NCT07377877
Title: Ultrasound-Guided External Oblique Intercostal Block Versus Erector Spinae Plane Block for Postoperative Analgesia After Laparoscopic Cholecystectomy: A Randomized Controlled Study
Brief Title: External Oblique Intercostal Block vs Erector Spinae Plane Block for Postoperative Analgesia After Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Elif Sarikaya Ozel, Principal Investigator- M.D. Karabuk Training and Research Hospital, Department of Anesthesiology, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOIBESP2026
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: External Oblique Intercostal Block; Erector Spina Plan Block; Pain Management
Keywords: External Oblique Intercostal Block; Erector Spinae Plane Block; Laparoscopic Cholecystectomy; Ultrasound-Guided Nerve Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either external oblique intercostal block or erector spinae plane block, and outcomes will be compared between two parallel intervention groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Block randomization lists will be generated using Microsoft Office 365 Excel (Microsoft, Redmond, WA, USA), and patients will be randomly assigned to one of the two study groups in a 1:1 ratio. According to the randomization result, group allocation will be placed in sealed opaque envelopes. Forty-five minutes before block performance, an independent nurse who is not involved in the study will deliver the envelope containing group assignment to the anesthesiologist performing the regional block.
  Patients, surgeons, ward nurses, and all personnel involved in postoperative data collection and outcome assessment will remain blinded to group allocation. Investigators responsible for outcome evaluation and statistical analysis will also be blinded to the randomization results.
  To ensure block quality and standardization, all regional blocks will be performed by a single experienced anesthesiologist who has performed each block technique at least 30 times. For masking purposes, this anesth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EOIB (Active Comparator): Patients allocated to the EOIB group will be transferred to the regional anesthesia area and monitored approximately 45 minutes before surgery. With the patient in the supine position, bilateral ultrasound-guided external oblique intercostal block (EOIB) will be performed. A total volume of 60 mL of 0.25% bupivacaine (30 mL per side) will be injected. General anesthesia will then be administered according to standard practice. In the postoperative period, additional analgesia will be provided using intravenous morphine patient-controlled analgesia (PCA).
  Interventions: Procedure: Ultrasound-Guided External Oblique Intercostal Block
- Group ESPB (Active Comparator): Patients allocated to the ESPB group will be transferred to the regional anesthesia area and monitored approximately 45 minutes before surgery. With the patient in the supine position, bilateral ultrasound-guided erector spinae plane block (ESPB) will be performed. A total volume of 60 mL of 0.25% bupivacaine (30 mL per side) will be injected. General anesthesia will then be administered according to standard practice. In the postoperative period, additional analgesia will be provided using intravenous morphine patient-controlled analgesia (PCA).
  Interventions: Procedure: Ultrasound-Guided Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Ultrasound-Guided External Oblique Intercostal Block — Bilateral ultrasound-guided external oblique intercostal block performed approximately 45 minutes before surgery. A total of 60 mL of 0.25% bupivacaine (30 mL per side) is injected into the fascial plane deep to the external oblique muscle.
  Arms: Group EOIB
Procedure: Ultrasound-Guided Erector Spinae Plane Block — Bilateral ultrasound-guided erector spinae plane block performed approximately 45 minutes before surgery. A total of 60 mL of 0.25% bupivacaine (30 mL per side) is injected into the fascial plane deep to the erector spinae muscle at the thoracic level under ultrasound guidance.
  Arms: Group ESPB

SUMMARY:
This randomized controlled study aims to compare the effects of the external oblique intercostal block (EOIB) and the erector spinae plane block (ESPB) on postoperative analgesia in adult patients undergoing elective laparoscopic cholecystectomy. Both EOIB and ESPB are ultrasound-guided regional anesthesia techniques currently used in clinical practice to improve postoperative pain control as part of multimodal analgesia strategies.

Laparoscopic cholecystectomy is a common minimally invasive surgical procedure; however, patients may still experience postoperative pain that can increase opioid consumption and delay recovery. Identifying the most effective regional anesthesia technique may improve postoperative analgesia and patient recovery.

In this study, eligible patients will be randomly assigned to receive either bilateral EOIB or bilateral ESPB in addition to standardized general anesthesia and postoperative patient-controlled analgesia. Postoperative pain scores, opioid consumption, quality of recovery, postoperative nausea and vomiting, and block-related complications will be evaluated during the first 24 hours after surgery. The study aims to provide comparative clinical evidence regarding the analgesic effectiveness of these two regional anesthesia techniques.

DETAILED DESCRIPTION:
This study is designed as a multicenter, prospective, randomized controlled trial aiming to evaluate and compare the postoperative analgesic outcomes of two ultrasound-guided regional anesthesia techniques, external oblique intercostal block (EOIB) and erector spinae plane block (ESPB), in adult patients undergoing elective laparoscopic cholecystectomy.EOIB and ESPB are ultrasound-guided regional anesthesia techniques that have been described for postoperative analgesia in upper abdominal surgery. In this study, the regional analgesic technique to be administered will be determined by randomization, while all other aspects of perioperative care will follow standard institutional practice. Except for the randomized allocation of the regional block technique, the research team will not alter routine anesthetic management.

The primary objective of the study is to compare cumulative intravenous morphine consumption during the first 24 hours after surgery between patients receiving EOIB and those receiving ESPB. Secondary objectives include assessment of postoperative pain scores at rest and during movement, quality of recovery, postoperative nausea and vomiting (PONV), intraoperative opioid consumption, rescue analgesic requirements, block-related complications, and opioid-related adverse effects.

Clinical Routine and Analgesic Protocol

All patients will be managed according to the standard multimodal analgesia protocol routinely used in the general surgery operating rooms of the participating institutions. Preoperatively, standard ASA monitoring will be applied, intravenous access will be established, and perioperative fluid management will be provided according to institutional practice. Mild sedation will be administered using intravenous midazolam at a dose of 0.02 mg/kg. Supplemental oxygen will be delivered via nasal cannula during block performance.

General anesthesia will be induced and maintained using routinely applied anesthetic agents. Intraoperative opioid administration will be titrated according to hemodynamic parameters to maintain mean arterial pressure and heart rate within acceptable limits, and total intraoperative opioid consumption will be recorded.

Postoperatively, all patients will receive intravenous paracetamol and intravenous tramadol as part of routine analgesic care. Intravenous morphine patient-controlled analgesia (PCA) will be provided to all patients using standardized settings, including a 1 mg bolus dose, a 10-minute lockout interval, and a 4-hour limit of 20 mg. Rescue analgesia will consist of intravenous tramadol infusion when pain remains uncontrolled (NRS ≥4), followed by intravenous morphine if necessary, according to the predefined protocol.

Block Techniques (Performed as Part of Study Protocol)

EOIB Group:

Patients allocated to the EOIB group will receive bilateral ultrasound-guided external oblique intercostal block approximately 45 minutes before surgery. With the patient in the supine position, a high-frequency linear ultrasound probe will be placed longitudinally along the anterior midaxillary line. Using an in-plane approach, a block needle will be advanced into the fascial plane deep to the external oblique muscle. A total volume of 30 mL of 0.25% bupivacaine will be administered bilaterally. The block will be performed by experienced anesthesiologists.

ESPB Group:

Patients allocated to the ESPB group will receive bilateral ultrasound-guided erector spinae plane block approximately 45 minutes before surgery. With the patient in the sitting position, following skin disinfection and sterile preparation, a convex ultrasound probe will be placed in a sagittal orientation approximately 2-3 cm lateral to the T7 spinous process. Using an in-plane approach, the needle will be advanced into the fascial plane deep to the erector spinae muscle. A total volume of 30 mL of 0.25% bupivacaine will be administered bilaterally, with sonographic confirmation of cranial and caudal spread.

Postoperative Assessment

Postoperative pain will be assessed using the 11-point Numeric Rating Scale (NRS; 0-10) at rest and during movement (deep breathing or coughing) at 0, 3, 6, 12, 18, and 24 hours after surgery. PONV will be evaluated using a verbal descriptive scale, and antiemetic treatment will be administered as needed according to institutional protocols.

Quality of recovery and patient satisfaction will be assessed using the Turkish version of the Quality of Recovery-15 (QoR-15) questionnaire at 24 hours postoperatively. Intraoperative opioid consumption, time to first PCA demand, rescue analgesic requirements, block-related complications (including pneumothorax, hematoma, vascular puncture, epidural spread, intrathecal injection, and local anesthetic systemic toxicity), and opioid-related side effects such as nausea, sedation, and respiratory depression will be recorded.

Dermatomal sensory block distribution will be assessed using a pinprick test with a 27-gauge needle 30 minutes after block application.

All data will be collected by trained personnel blinded to group allocation. Due to the low-risk nature of the interventions and the short follow-up period, no independent data monitoring committee has been established.

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 80 years
* Scheduled to undergo elective laparoscopic cholecystectomy
* Classified as American Society of Anesthesiologists (ASA) physical status I-III
* Ability to understand and operate a patient-controlled analgesia (PCA) device
* Provision of written informed consent

Exclusion Criteria

* History of chronic opioid use for more than four weeks prior to surgery
* Presence of pre-existing chronic pain conditions, such as migraine or fibromyalgia
* History of alcohol or substance abuse
* Known hypersensitivity or allergy to local anesthetics or opioids
* Presence of severe organ dysfunction, including clinically significant hepatic or renal disease
* Any contraindication to regional anesthesia
* Severe psychiatric disorders impairing patient cooperation or the ability to reliably assess pain (e.g., psychosis, dementia)
* Pregnancy or breastfeeding
* Presence of hematological disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
24-hour cumulative opioid consumption | postoperative day 1
  Total opioid consumption within the first 24 hours, including PCA-administered morphine and rescue analgesics converted to morphine milligram equivalents (MME).

SECONDARY OUTCOMES:
12-hour cumulative opioid consumption | postoperative 12th hour
  Total opioid consumption within the first 12 hours, including PCA-administered morphine and rescue analgesics converted to MME.
Postoperative pain scores (NRS at rest) | postoperative day 1
  Pain status at rest will be assessed by numeric rating scale (NRS) score at 0, 3, 6, 12, 18 and 24 hours after surgery. In addition, the time until the first analgesic requirement will be recorded. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Postoperative pain scores (NRS during activity) | postoperative day 1
  Pain status during activity will be assessed by numeric rating scale (NRS) score at 0, 3, 6, 12, 18 and 24 hours after surgery. In addition, the time until the first analgesic requirement will be recorded. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Patient-reported quality of recovery (QoR-15 score) | postoperative day 1
  Quality of recovery will be assessed using the validated 15-item Quality of Recovery questionnaire (QoR-15). Each item is scored on an 11-point numeric scale (0-10), resulting in a total score ranging from 0 to 150, with higher scores indicating better postoperative recovery.
Postoperative nausea and vomiting incidence (PONV) | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18 and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required (The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once).
Time to first PCA analgesic demand | Postoperative day 1
  Time at which the first analgesic is requested
Number of patients requiring rescue analgesia | Postoperative day 1
  The number of patients requiring rescue analgesia due to inadequate postoperative pain control (Numeric Rating Scale [NRS] ≥4) despite standard analgesic management
Block-related complications | Postoperative day 7
  Incidence of complications such as bleeding, hematoma, or local anesthetic systemic toxicity (LAST)
Opioid-related adverse effects | Postoperative day 7
  Presence of itching, sedation, fatigue, or respiratory depression related to opioid use.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Sarikaya Ozel, M.D., Principal Investigator — Karabuk Training and Research Hospital, Department of Anesthesiology
Locations (2):
- Turkey (Türkiye) (2):
  - Karabuk Training and Research Hospital, Department of Anesthesiology and Reanimation, Karabük
  - Department of Anesthesiology and Reanimation, Samsun City Hospital, Samsun

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team, as the dataset contains sensitive clinical information and data sharing was not included in the original informed consent. Data will be used solely for the purposes of the current study and related scientific publications, in accordance with institutional policies and ethical regulations.